CLINICAL TRIAL: NCT02088138
Title: Effects of Functional Electrical Stimulation on Physical Performance of Patients in Cardiac Rehabilitation
Brief Title: Functional Electrical Stimulation in Cardiac Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Antônio Marcos Vargas da Silva (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Antônio Marcos Vargas da Silva, PhD in Physiology, Universidade Federal de Santa Maria
Organization: Universidade Federal de Santa Maria (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FESCP01
Record Dates: First submitted 2014-02-26; First posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Coronary Disease; Heart Failure
Keywords: Thoracic Surgery; Electrical Stimulation; Rehabilitation; Quality of Life
MeSH Terms: conditions — Coronary Disease; Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Functional Electrical Stimulation (Experimental): Functional Electrical Stimulation
  In the intervention group the FES was applied in the medial and lateral vastus of both thighs targeting the movement of knee extension. The application frequency was 15 Hz, lasting 40 minutes, pulse width of 0.5 ms, time ON 5s, time OFF 10s, ramp-up of 0 or 1s, descent ramp 2s and intensity as tolerance patient.
  Interventions: Device: Functional Electrical Stimulation
- FES placebo (Experimental): Functional Electrical Stimulation placebo
  The placebo group received functional electrical stimulation with the same parameters in the intervention group, except that the intensity of stimulation did not lead to visible or palpable contraction.
  Interventions: Device: Functional Electrical Stimulation placebo

INTERVENTIONS:
Device: Functional Electrical Stimulation — Functional electrical stimulation twice per week for eight weeks totaling sixteen sessions.
  Other Names: FES
  Arms: Functional Electrical Stimulation
Device: Functional Electrical Stimulation placebo — Functional electrical stimulation in the sensory threshold level, twice a week for eight weeks, totaling sixteen sessions.
  Other Names: FES placebo
  Arms: FES placebo

SUMMARY:
The purpose of this study was to determine the effects of Functional Electrical Stimulation (FES) on physical performance and quality of life of patients in cardiac rehabilitation.

DETAILED DESCRIPTION:
This randomized controlled trial aimed to evaluate the effects of functional electrical stimulation (FES) in patients with stage II and III cardiac rehabilitation (CR) on the variables strength, endurance and muscle tropism lower limb, functional capacity and quality of life. To this were invited to participate in the study cardiac patients registered in the database of the cardiology department of the University Hospital of Santa Maria. The sample included patients of both sexes undergoing coronary artery bypass grafting or valve replacement. The subjects were divided into two groups: placebo group (PG) or functional electrical stimulation group (FESG). To verify the effect of this intervention, before and after the protocol patients underwent the following evaluations: one repetition maximum test, sit-and-stand test, perimetry thighs, the six-minute walk test and evaluate the quality of life through The Medical questionnaire Study 36-item Short-Form Health Survey (SF-36).

ELIGIBILITY:
Inclusion Criteria:

* Patients in phase II and III of cardiac rehabilitation undergoing coronary artery bypass grafting or valve replacement

Exclusion Criteria:

* Patients with some cognitive impairment that prevents the completion of assessments, inability to understand the term of free and informed consent or with the following contraindications to the use of FES: epidermal lesions at the site of application, change of skin sensitivity or intolerance electrical stimulator;
* Patients undergoing cardiac surgery other than coronary artery bypass grafting or valve replacement;
* Patients who use pacemakers;
* Subjects with peripheral vascular changes in the lower limbs;
* Presence of comorbidities such as chronic obstructive pulmonary disease (COPD), cerebrovascular disease or skeletal muscle disease.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Distance on the six minute walk test | Two Years

SECONDARY OUTCOMES:
Lower limb muscle strength measured by the load (kg) sustained in one repetition maximum test | Two years
Quality of life through The Medical Study 36-Item Short-Form Health Survey (SF-36) questionnaire | Two years
Lower limb muscle tropism evaluated by measuring the thigh circumference by tape | Two years
Lower limb muscle endurance assessed by sit-and-stand test | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Antônio M Vargas da Silva, PhD, Principal Investigator — Universidade Federal de Santa Maria
Locations (3):
- Brazil (3):
  - Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Federal University of Santa Maria, Santa Maria, Rio Grande do Sul